CLINICAL TRIAL: NCT05847699
Title: Radiohistological Correlation of Thrombohemorrhagic Remodeling in the Acute Phase of Ischemic Stroke Managed by Decompressive Hemicraniectomy
Acronym: SWI-SURGERY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: JDS_2023_1
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient intervention (Other): Patients who need to undergo an MRI prior to a possible decompressive hemicraniectomy (DH) as part of the treatment of an acute ischemic stroke.
  Or Patients who have undergone a post-thrombectomy brain scan and are indicated for a possible decompressive hemicraniectomy as part of the treatment of an acute ischemic stroke.
  Interventions: Other: MRI sequences and biopsies

INTERVENTIONS:
Other: MRI sequences and biopsies — Addition of a contrast injection and optimized SWI sequences during the pre-DH MRI examination performed as part of the care Addition of two 1x1 cm biopsy samples of cortex in two different non-functional ischemic areas, one of which is within the SWI hyposignal remodeling, during the DH. This will be a cold pial dissection without the use of coagulation.

SUMMARY:
Recent years have witnessed a change in the therapeutic paradigm of stroke with the advent of mechanical thrombectomy as the reference treatment.

However, despite the achievement of effective proximal recanalization in nearly 80% of patients, nearly half of these patients have an unfavorable functional outcome. Several causes can be mentioned, such as the extent of the initial ischemic damage, the occurrence of complications related to reperfusion treatments or the occurrence of thrombosis of the downstream microvascularization. The latter is a phenomenon that has been known and studied increasingly over the last twenty years. It is the result of multiple cellular remodeling following ischemia and at the origin of an endoluminal filling by platelets, inflammatory cells and fibrin. This phenomenon introduces the fundamental difference between recanalization, i.e. the removal of the obstruction by the thrombus, and reperfusion, which translates into a satisfactory supply of oxygen to the ischemic tissues and therefore the expected result of these treatments. However, not all recanalization is necessarily accompanied by reperfusion, which is the phenomenon of no-reflow. This last situation could be explained by downstream microvascular thrombosis. Studies have shown the interest of intravenous thrombolysis associated with mechanical thrombectomy to preserve this vascular bed and improve cerebral reperfusion. More recently, a study has also shown the value of adding intra-arterial thrombolysis after mechanical thrombectomy. Nevertheless, there is currently no clinical evidence of the reality and prognostic importance of downstream microvascular thrombosis.

Advances in imaging have allowed the development of susceptibility weighted imaging (SWI) sequences with millimeter resolution, allowing a precise study of vascular damage and the appearance of previously unseen remodeling. Among them, the existence of cortical or juxta-cortical microinfarcts whose remnographic characteristics differed by the presence of a SWI hyposignal. The hypothesis evoked is that of a hemorrhagic remodeling consecutive to the barrier rupture. However, in view of the pathophysiology explained so far and the hypointense character of the thrombi on the SWI sequences, these remodeling could in fact be not microbleeding but rather markers of thrombosis in the downstream microcirculation. MRI would allow to identify the presence and the importance of microvascular thrombosis and thus to bring arguments to specifically target this microvascular component, consequence of cerebral ischemia, by antithrombotic or thrombolytic treatments.

The objective of our project is therefore to carry out a study focused on a better description and understanding of cortical and basal ganglia SWI hyposignals with a histopathological correlation and with the clinical prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Managed for sylvian ischemic stroke
* Requiring brain MRI as part of the evaluation for possible decompressive hemicraniectomy (DH).

Or

* Having undergone a post-thrombectomy brain scan showing cortical hyperdensities and indication for a possible decompressive hemicraniectomy
* Consent to participate in the study
* Affiliated or beneficiary of a health insurance plan

Exclusion Criteria:

* Absolute or relative contraindication to gadobutrol injection (history of true allergic reaction or intolerance to gadobutrol, renal insufficiency with creatinine clearance <15ml/min). In particular, if an allergic reaction was observed during the injection of gadobutrol performed for care during the acute phase MRI a few hours or days before.
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2028-10-02 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare the amount of microvascular thrombosis between samples taken in areas of SWI hyposignal on MRI and those taken in SWI isosignal areas. | Day 0
  Vascular microthrombosis defined as % of vessels affected/mm2

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, France